CLINICAL TRIAL: NCT00768404
Title: A Phase I, Open-Label, Parallel-Group, Single Dose, Non-Randomized Study To Compare The Pharmacokinetics Of Each Individual Component (Topiramate And Phentermine) Of The Combination Product VI-0521 In Subjects With Mild, Moderate And Severe Renal Impairment To Subjects With Normal Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics of VI-0521 Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OB-106
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Phentermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Topirmate and Phentermine

INTERVENTIONS:
Drug: Topirmate and Phentermine — A single oral dose of the combination product VI-0521 (15 mg phentermine and 92 mg topiramate) will be administered with 240 mL of water at hour 0.

SUMMARY:
VI-0521, a fixed dose combination of immediate-release (IR) phentermine and controlled-release (CR) topiramate, is in Phase III clinical development as a potential therapy for obesity. In human, both phentermine and topiramate are primarily cleared by renal excretion. The contribution of hepatic metabolism to elimination of phentermine and topiramate is not significant. Obese patients, the proposed indicated population for future treatment with VI-0521, are likely to have renal impairment. Therefore, this study is important in understanding the effect of renal impairment on the pharmacokinetics of topiramate and phentermine in subjects with renal impairment compared to subjects with normal renal function.

DETAILED DESCRIPTION:
This open-label, parallel-group, single dose, non-randomized study will be conducted at multiple sites in the United States in which up to 40 male and female subjects, 19-75 years of age (inclusive), with varying degrees of renal function may be enrolled and dosed to obtain at least 32 evaluable subjects (4 groups, 8 subjects per group). Subjects will report to the study site on the evening before treatment and will remain at the site until the 48-hour PK sample has been drawn (approximately 3 days). All subjects will be fasted overnight for a minimum of 8 hours before drug treatment in the morning. A single oral dose of the combination product VI-0521 (15 mg phentermine and 92 mg topiramate) will be administered with 240 mL of water at hour 0. Standard meals will be provided uniformly to all subjects at approximately 4 and 9 hours after dosing, and an evening snack will be provided approximately 12 - 13 hours after dosing. Blood samples for the determination of phentermine and topiramate concentrations in plasma will be collected at 0 (pre-dose), 1, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 36 and 48 hours post dosing. Subjects will be released from the study site following the 48-hour sample but will return to the site for PK sampling at 72, 96, 120, 144, 168 and 192 hours post dose. The severe renal impairment group will be given the option to stay at the site for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

Group 1 will consist of 8-10 males or females with normal renal function, 19-75 years of age, inclusive.

Groups 2-4 will consist of 8-10 males or females per group with varying degree of stable renal impairment

Exclusion Criteria:

A history or presence of significant cardiovascular, neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the investigator; any history of glaucoma, increased intraocular pressure, or medications to treat increased intraocular pressure; presence of cholelithiasis or cholecystitis within the last 6 months that has not been surgically treated with cholecystectomy; any history of a cardiovascular or cerebrovascular event; subjects requiring dialysis; any active malignancy except basal cell carcinoma; systolic blood pressure > 180 mm Hg or diastolic blood pressure > 100 mm Hg at screening or at check-in (2 rechecks are allowed); Hemoglobin <12.0 g/dL for Group 1 (patients with normal renal function); Hemoglobin <. 9.0 g/dL for Groups 2, 3 and 4 (patients with mild to severe renal function) positive drug/alcohol test at screening or check in; blood donation or significant blood loss within 56 days of dosing; plasma donation within 7 days of dosing. In female subjects, a positive pregnancy test at screening or check-in is exclusionary

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC
Locations (4):
- United States (4):
  - Advanced Clinical Research Institute, Anaheim, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota